CLINICAL TRIAL: NCT00404651
Title: Lot to Lot Consistency Study of DTaP-IPV-Hep B-PRP~T Vaccine Administered at 2-4-6 Months of Age in Healthy Mexican Infants
Brief Title: Lot Consistency Study of DTaP-IPV-HB-PRP~T Vaccine Administered at 2-4-6 Months of Age in Healthy Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: A3L11
Record Dates: First submitted 2006-11-28; First posted 2006-11-29 (Estimated); Results first posted 2014-05-09 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-04

CONDITIONS: Diphtheria; Tetanus; Pertussis; Hepatitis B; Poliomyelitis
Keywords: Diphtheria; Tetanus; Pertussis; Hepatitis B; Poliomyelitis; Invasive Haemophilus influenzae type b.
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Hepatitis B; Poliomyelitis | interventions — DTaP-IPV-HB-PRP-T vaccine; diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 (Experimental): Participants receive vaccine Batch A
  Interventions: Biological: DTaP-IPV-HB-PRP~T vaccine
- Group 2 (Experimental): Participants receive vaccine Batch B
  Interventions: Biological: DTaP-IPV-HB-PRP~T vaccine
- Group 3 (Experimental): Participants receive vaccine Batch C
  Interventions: Biological: DTaP-IPV-HB-PRP~T vaccine
- Group 4 (Active Comparator): Participants receive Infanrix hexa™
  Interventions: Biological: DTaP-HBV-IPV vaccine

INTERVENTIONS:
Biological: DTaP-IPV-HB-PRP~T vaccine — 0.5 mL, intramuscular (IM)
  Arms: Group 1
Biological: DTaP-IPV-HB-PRP~T vaccine — 0.5 mL, IM
  Arms: Group 2
Biological: DTaP-IPV-HB-PRP~T vaccine — 0.5 mL, IM
  Arms: Group 3
Biological: DTaP-HBV-IPV vaccine — 0.5 mL, IM
  Other Names: INFANRIX®HEXA
  Arms: Group 4

SUMMARY:
The purpose of this trial is to clinically confirm that the manufacturing process of the final bulk products of the investigational DTaP-IPV-HB-PRP~T vaccine is consistent.

The primary objective is to demonstrate the equivalence of three batches of DTaP-IPV-HB-PRP~T vaccine, in terms of seroprotection and seroconversion rates for the vaccine antigens after the three-dose primary series.

The secondary objectives are:

* To describe in each group, the immunogenicity parameters for all antigens one month after the third dose of the primary series
* To assess the overall safety in each group one month after the third dose of the primary series.

ELIGIBILITY:
Inclusion Criteria :

* Two months old infants on the day of inclusion
* Born at full term of pregnancy (≥ 37 weeks) with a birth weight ≥ 2.5 kg
* Informed consent form signed by one or both parents or by the guardian and two independent witnesses
* Able to attend all scheduled visits and to comply with all trial procedures
* Received Bacillus Calmette Guerin (BCG) vaccine between birth and one month of life in agreement with the national immunization calendar.

Exclusion Criteria :

* Participation in another clinical trial in the four weeks preceding the (first) trial vaccination
* Planned participation in another clinical trial during the present trial period
* Congenital or acquired immunodeficiency
* Systemic hypersensitivity to any of the vaccine components or history of a life-threatening reaction to the trial vaccine or a vaccine containing the same substances
* Chronic illness at a stage that could interfere with trial conduct or completion
* Blood or blood-derived products received since birth
* Any vaccination in the four weeks preceding the first trial visit
* Any planned vaccination (except BCG, rotavirus, and pneumococcal conjugated vaccines) during the study
* Documented history of pertussis, tetanus, diphtheria, poliomyelitis, Haemophilus influenzae type b or hepatitis B infection(s) (confirmed either clinically, serologically or microbiologically)
* Previous vaccination against hepatitis B, pertussis, tetanus, diphtheria, poliovirus, or Haemophilus influenzae type b infection(s)
* Known personal or maternal history of HIV, Hepatitis B (HBsAg) or Hepatitis C seropositivity
* Thrombocytopenia or a bleeding disorder contraindicating intramuscular vaccination
* History of seizures
* Febrile (rectal equivalent temperature ≥ 38.0°C) or acute illness on the day of inclusion.

Min Age: 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1189 (Actual)
Dates: Start 2006-11; Primary Completion 2008-04 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (5):
- Mexico (5):
  - Estado de México
  - Insurgentes Cuicuilco
  - Monterrey
  - Puebla City
  - Tlalpan

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 14 November 2006 to 13 July 2007 in 6 clinical centers in Mexico.
Pre-assignment Details: A total of 1189 participants who met the inclusion and exclusion criteria were enrolled and vaccinated.
Groups:
- DTaP-IPV-HB-PRP~T Batch 1: Participants received 3 doses of Batch 1 of diphtheria (D), tetanus (T), pertussis (2 component acellular), recombinant hepatitis B Hansenula (Hep B) and poliomyelitis (IPV) vaccine adsorbed, and Haemophilus influenzae type b (Hib) vaccine, conjugated to tetanus protein (DTaP-IPV-Hep B-PRP~T), with one dose each at 2, 4, and 6 months of age.
- DTaP-IPV-HB-PRP~T Batch 2: Participants received 3 doses of Batch 2 of diphtheria (D), tetanus (T), pertussis (2 component acellular), recombinant hepatitis B Hansenula (Hep B) and poliomyelitis (IPV) vaccine adsorbed, and Haemophilus influenzae type b (Hib) vaccine, conjugated to tetanus protein (DTaP-IPV-HB-PRP~T), with one dose each at 2, 4, and 6 months of age.
- DTaP-IPV-HB-PRP~T Batch 3: Participants received 3 doses of Batch 3 of diphtheria (D), tetanus (T), pertussis (2 component acellular), recombinant hepatitis B Hansenula (Hep B) and poliomyelitis (IPV) vaccine adsorbed, and Haemophilus influenzae type b (Hib) vaccine, conjugated to tetanus protein (DTaP-IPV-HB-PRP~T), with one dose each at 2, 4, and 6 months of age.
- Infanrix Hexa™: Participants received 3 doses of diphtheria (D), tetanus (T), pertussis (2 component acellular), recombinant hepatitis B Hansenula (Hep B) and poliomyelitis (IPV) vaccine adsorbed (Infanrix hexa™), plus Haemophilus influenzae type b (Hib) vaccine conjugated to tetanus protein , with one dose each at 2, 4, and 6 months of age.
Period: Overall Study
Arm/Group | DTaP-IPV-HB-PRP~T Batch 1 | DTaP-IPV-HB-PRP~T Batch 2 | DTaP-IPV-HB-PRP~T Batch 3 | Infanrix Hexa™
Started | 340 | 343 | 339 | 167
Completed | 301 | 315 | 294 | 146
Not Completed | 39 | 28 | 45 | 21
Not completed — Serious Adverse Event | 0 | 0 | 2 | 0
Not completed — Protocol Violation | 10 | 5 | 14 | 5
Not completed — Lost to Follow-up | 15 | 11 | 13 | 10
Not completed — Withdrawal by Subject | 14 | 12 | 16 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DTaP-IPV-HB-PRP~T Batch 1 | DTaP-IPV-HB-PRP~T Batch 2 | DTaP-IPV-HB-PRP~T Batch 3 | Infanrix Hexa™ | Total
Number analyzed (Participants) | 340 | 343 | 339 | 167 | 1189
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 340 | 343 | 339 | 167 | 1189
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Months] | 2.00 (0.200) | 2.00 (0.197) | 2.01 (0.193) | 1.98 (0.189) | 2.00 (0.195)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 160 | 163 | 167 | 82 | 572
  Male | 180 | 180 | 172 | 85 | 617
Region of Enrollment [Number; unit: Participants]
  Mexico | 340 | 343 | 339 | 167 | 1189

OUTCOME MEASURES:

1. Primary Outcome: Equivalence of Seroprotection Against Vaccine Antigens in Study Participants After Vaccination With Either One of the Batches of DTaP-IPV-HB-PRP~T or Infanrix Hexa™ Vaccine
Description: Antibody titers were measured for hepatitis B (Hep B) by enhanced chemiluminescence detection, for Haemophilus influenzae type b (PRP) by Farr type radioimmunoassay, for Diphtheria (D) by toxin neutralization test, and for Tetanus (T) by enzyme-linked immunosorbent assay (ELISA). Seroprotection was defined as a titer ≥ 0.10 mIU/mL for Hep B, ≥ 0.15 µg/mL for PRP, and ≥ 0.01 IU/mL for D and T antibodies.
Time Frame: Day 150 (one month post-dose 3)
Population: Seroprotection was assessed in participants that received a vaccine who did not have any protocol deviation that might have interfered with primary criteria evaluation (Per-Protocol Population). Total number (N) are those with available data for the endpoint.
Measure: Number; unit: Participants
Arm/Group | DTaP-IPV-HB-PRP~T Batch 1 | DTaP-IPV-HB-PRP~T Batch 2 | DTaP-IPV-HB-PRP~T Batch 3 | Infanrix Hexa™
Number analyzed (Participants) | 231 | 236 | 228 | 119
Participants
  Anti-Hep B (N = 230, 234, 236, 119) | 226 | 231 [0 to 0] | 221 [0 to 0] | 119 [0 to 0]
  Anti-PRP (N = 231, 236, 228, 119) | 229 | 232 [0 to 0] | 226 [0 to 0] | 118 [0 to 0]
  Anti-Diphtheria (N = 231, 236, 228, 119) | 220 | 228 [0 to 0] | 222 [0 to 0] | 118 [0 to 0]
  Anti-Tetanus (N = 231, 236, 227, 119) | 231 | 236 [0 to 0] | 227 [0 to 0] | 119 [0 to 0]

2. Primary Outcome: Equivalence of Seroprotection Against Pertussis in Study Participants After Vaccination With Either One of the Batches of DTaP-IPV-HB-PRP~T or Infanrix Hexa™ Vaccine.
Description: Antibody titers were measured for pertussis toxoid (PT) and filamentous hemagglutinin (FHA) by enzyme linked immunosorbent assay (ELISA). Seroconversion was defined as a ≥ 4 fold increase in titer from Day 0 (before dose 1) to Day 150, one month post-dose 3.
Time Frame: Day 150 (one month post-dose 3)
Population: Seroconversion was assessed in all participants who did not have any protocol deviation that might have interfered with primary criteria evaluation (Per-Protocol Population).
Measure: Number; unit: Participants
Arm/Group | DTaP-IPV-HB-PRP~T Batch 1 | DTaP-IPV-HB-PRP~T Batch 2 | DTaP-IPV-HB-PRP~T Batch 3 | Infanrix Hexa™
Number analyzed (Participants) | 231 | 236 | 228 | 119
Participants
  Anti-Pertussis (N= 228, 234, 223, 118) | 223 | 226 [0 to 0] | 218 [0 to 0] | 113 [0 to 0]
  Anti-FHA (N= 227, 233, 221, 115) | 225 | 229 [0 to 0] | 216 [0 to 0] | 111 [0 to 0]

3. Primary Outcome: Equivalence of Seroprotection Against Poliovirus Types 1, 2, and 3 in Study Participants After Vaccination With Either One of the Batches of DTaP-IPV-Hep B-PRP~T or Infanrix Hexa™ Vaccine
Description: Antibody titers were measured for poliovirus types 1, 2, and 3 by Enzyme immuno assay. Seroprotection against Poliovirus Types 1, 2, and 3 was defined as a titer ≥ 8 (1/dilutions).
Time Frame: Day 150 (one month post-dose 3)
Population: Seroprotection was assessed in all participants who did not have any protocol deviation that might have interfered with primary criteria evaluation (Per-Protocol Population).
Measure: Number; unit: Participants
Arm/Group | DTaP-IPV-HB-PRP~T Batch 1 | DTaP-IPV-HB-PRP~T Batch 2 | DTaP-IPV-HB-PRP~T Batch 3 | Infanrix Hexa™
Number analyzed (Participants) | 231 | 236 | 228 | 119
Participants
  Anti-Polio 1 (N = 231, 236, 225, 119) | 230 | 236 [0 to 0] | 225 [0 to 0] | 119 [0 to 0]
  Anti-Polio 2 (N = 230, 236, 226, 118) | 230 | 236 [0 to 0] | 226 [0 to 0] | 118 [0 to 0]
  Anti-Polio 3 (N = 230, 236, 226, 119) | 229 | 235 [0 to 0] | 226 [0 to 0] | 117 [0 to 0]

4. Secondary Outcome: Geometric Mean Titers of Antibodies After Vaccination With Either One of the Batches of DTaP-IPV-HB-PRP~T Vaccine or Infanrix Hexa™ Vaccine
Description: Antibody titers were measured for hepatitis B (Hep B) by enhanced chemiluminescence detection, for Haemophilus influenzae type b (PRP) by Farr type radioimmunoassay, for diphtheria (D) by toxin neutralization test, and for tetanus by enzyme linked immunosorbent assay. Antibody titers were measured for poliovirus types 1, 2, and 3 by neutralization assay. Antibody titers were measured for pertussis toxoid (PT) and filamentous hemagglutinin (FHA) by enzyme linked immunosorbent assay (ELISA).
Time Frame: Day 150 (one month post-dose 3)
Population: Geometric Mean Titers were assessed in all participants with endpoint data who did not have any protocol deviation that might have interfered with primary criteria evaluation (Per-Protocol Population).
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | DTaP-IPV-HB-PRP~T Batch 1 | DTaP-IPV-HB-PRP~T Batch 2 | DTaP-IPV-HB-PRP~T Batch 3 | Infanrix Hexa™
Number analyzed (Participants) | 231 | 236 | 228 | 119
Titers
  Anti-Hep B (N = 230, 234, 226, 119) | 935 [755 to 1158] | 1566 [1288 to 1905] | 1009 [814 to 1252] | 1576 [1283 to 1934]
  Anti-PRP (N = 231, 236, 228, 119) | 11.9 [9.77 to 14.5] | 13.1 [10.7 to 16.0] | 11.5 [9.26 to 14.3] | 6.68 [5.10 to 8.74]
  Anti-Diphtheria (N = 231, 236, 228, 119) | 0.176 [0.143 to 0.217] | 0.246 [0.194 to 0.311] | 0.173 [0.139 to 0.214] | 0.173 [0.132 to 0.226]
  Anti-Tetanus (N = 231, 236, 227, 119) | 1.90 [1.67 to 2.15] | 1.86 [1.64 to 2.10] | 1.77 [1.57 to 2.01] | 2.20 [1.93 to 2.52]
  Anti-Polio 1 (N = 231, 236, 225, 119) | 860 [725 to 1021] | 945 [809 to 1102] | 843 [712 to 999] | 1370 [1082 to 1736]
  Anti-Polio 2 (N = 230, 236, 226, 118) | 1689 [1429 to 1996] | 1665 [1416 to 1957] | 1612 [1374 to 1892] | 2337 [1878 to 2909]
  Anti-Polio 3 (N = 230, 235, 226, 117) | 1198 [1015 to 1413] | 1170 [995 to 1377] | 962 [809 to 1143] | 2186 [1752 to 2727]
  Anti-Pertusiss toxoid (N = 230, 235, 226, 119) | 242 [226 to 260] | 238 [220 to 258] | 241 [222 to 262] | 228 [205 to 254]
  Anti-FHA (N = 230, 234, 226, 118) | 243 [228 to 259] | 256 [237 to 277] | 220 [202 to 239] | 182 [165 to 200]

5. Secondary Outcome: Number of Participants Reporting Solicited Injection Site or Systemic Reactions After Vaccination With Either One of the Batches of DTaP-IPV-HB-PRP~T Vaccine or Infanrix Hexa™ Vaccine
Description: Solicited Injection Site Reactions: Pain, Erythema, and Swelling. Solicited Systemic Reactions: Fever ([pyrexia] - temperature), Vomiting, Crying, Somnolence, Anorexia, and Irritability
Time Frame: Day 0 (pre-each vaccination) up to 7 days post-each dose
Population: Solicited reactions were assessed in all subjects who received at least one dose of vaccine, according to the vaccine actually received (Safety Analysis Population). Two batch 1 subjects got batch 2 vaccine, and 1 batch 1 got batch 3 vaccine. Total number (N) are those with available data for the outcome
Measure: Number; unit: Participants
Arm/Group | DTaP-IPV-HB-PRP~T Batch 1 | DTaP-IPV-HB-PRP~T Batch 2 | DTaP-IPV-HB-PRP~T Batch 3 | Infanrix Hexa™
Number analyzed (Participants) | 337 | 345 | 340 | 167
Participants
  Pain Post-dose 1 (N = 323, 336, 329, 155) | 220 | 237 [0 to 0] | 225 [0 to 0] | 95 [0 to 0]
  Pain Post-dose 2 (N = 310, 319, 316, 153) | 191 | 220 [0 to 0] | 199 [0 to 0] | 88 [0 to 0]
  Pain Pos-dose 3 (N = 302, 317, 306, 149) | 188 | 209 [0 to 0] | 198 [0 to 0] | 87 [0 to 0]
  Erythema-Post dose 1 (N = 323, 336, 329, 156) | 92 | 97 [0 to 0] | 97 [0 to 0] | 41 [0 to 0]
  Erythema Post-dose 2 (N = 310, 319, 315, 153) | 94 | 101 [0 to 0] | 96 [0 to 0] | 33 [0 to 0]
  Erythema Post-dose 3 (N = 302, 317, 306, 149) | 95 | 94 [0 to 0] | 101 [0 to 0] | 43 [0 to 0]
  Swelling Post-dose 1 (N = 323, 336, 329, 156) | 67 | 86 [0 to 0] | 80 [0 to 0] | 35 [0 to 0]
  Swelling Post-dose 2 (N = 310, 319, 315, 153) | 74 | 70 [0 to 0] | 60 [0 to 0] | 26 [0 to 0]
  Swelling Post-dose 3 (N = 302, 317, 306, 149) | 66 | 65 [0 to 0] | 72 [0 to 0] | 22 [0 to 0]
  Pyrexia Post-dose 1 (N = 323, 336, 329, 156) | 63 | 77 [0 to 0] | 82 [0 to 0] | 17 [0 to 0]
  Pyrexia Post-dose 2 (N = 310, 318, 315, 153) | 75 | 84 [0 to 0] | 85 [0 to 0] | 32 [0 to 0]
  Pyrexia Post-dose 3 (N = 302, 317, 306, 149) | 69 | 85 [0 to 0] | 70 [0 to 0] | 28 [0 to 0]
  Vomiting Post-dose 1 (N = 323, 336, 329, 156) | 68 | 63 [0 to 0] | 56 [0 to 0] | 27 [0 to 0]
  Vomiting Post-dose 2 (N = 310, 319, 316, 153) | 37 | 46 [0 to 0] | 34 [0 to 0] | 18 [0 to 0]
  Vomiting Post-dose 3 (N = 302, 317, 306, 149) | 51 | 46 [0 to 0] | 47 [0 to 0] | 20 [0 to 0]
  Crying Post-dose 1 (N = 323, 336, 329, 156) | 160 | 156 [0 to 0] | 148 [0 to 0] | 62 [0 to 0]
  Crying Post-dose 2 (N=310, 319, 316, 153) | 133 | 145 [0 to 0] | 134 [0 to 0] | 59 [0 to 0]
  Crying Post-dose 3 (N=302, 317, 306, 149) | 110 | 118 [0 to 0] | 122 [0 to 0] | 40 [0 to 0]
  Somnolence Post-dose 1 (N = 323, 336, 329, 156) | 93 | 110 [0 to 0] | 102 [0 to 0] | 45 [0 to 0]
  Somnolence Post-dse 2 (N = 310, 319, 316, 153) | 69 | 78 [0 to 0] | 65 [0 to 0] | 24 [0 to 0]
  Somnolence Post-dose 3 (N = 302, 317, 306, 149) | 56 | 57 [0 to 0] | 54 [0 to 0] | 20 [0 to 0]
  Anorexia Post-dose 1 (N = 323, 336, 329, 156) | 62 | 75 [0 to 0] | 70 [0 to 0] | 27 [0 to 0]
  Anorexia Post-dose 2 (N = 310, 319, 315, 153) | 56 | 64 [0 to 0] | 65 [0 to 0] | 25 [0 to 0]
  Anorexia Post-dose 3 (N = 302, 317, 306, 149) | 61 | 58 [0 to 0] | 65 [0 to 0] | 29 [0 to 0]
  Irritability Post-dose 1 (N = 323, 336, 329, 156) | 188 | 198 [0 to 0] | 193 [0 to 0] | 83 [0 to 0]
  Irritability Post-dose 2 (N = 310, 319, 316, 153) | 158 | 192 [0 to 0] | 174 [0 to 0] | 72 [0 to 0]
  Irritability Post-dse 3 (N = 302, 317, 306, 149) | 158 | 167 [0 to 0] | 165 [0 to 0] | 69 [0 to 0]

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from Day 0 after the first vaccination for up to 10 months (Day 300) post-vaccination.
Description: Safety was assessed in all participants who received at least one dose of vaccine, according to the vaccine actually received (Safety Analysis Population). Two participants randomized to Batch 1 got Batch 2 vaccine; 1 Batch 1 participant got Batch 3 vaccine. Total number (N) for each safety parameter are those with available data.
Arm/Group | DTaP-IPV-HB-PRP~T Batch 1 | DTaP-IPV-HB-PRP~T Batch 2 | DTaP-IPV-HB-PRP~T Batch 3 | Infanrix Hexa™
Serious Adverse Events (participants affected / at risk) | 5/337 | 5/345 | 12/340 | 6/167
Other Adverse Events (participants affected / at risk) | 220/337 | 237/345 | 225/340 | 95/167
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DTaP-IPV-HB-PRP~T Batch 1 (N=337) | DTaP-IPV-HB-PRP~T Batch 2 (N=345) | DTaP-IPV-HB-PRP~T Batch 3 (N=340) | Infanrix Hexa™ (N=167)
Heart Disease Congenital (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intussusception (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Bronchopneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 2 (2) | 5 (5) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multiple Fractures (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Food Intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile Convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 1 (2) | 1 (1)
Infantile Spasms (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Partial Seizures (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | DTaP-IPV-HB-PRP~T Batch 1 (N=337) | DTaP-IPV-HB-PRP~T Batch 2 (N=345) | DTaP-IPV-HB-PRP~T Batch 3 (N=340) | Infanrix Hexa™ (N=167)
Vomiting (Gastrointestinal disorders) | 68/323 (68) | 63/336 (63) | 56/329 (56) | 27/156 (27)
Injection Site Pain (General disorders) | 220/323 (220) | 237/336 (237) | 225/329 (225) | 95/155 (95)
Injection Site Erythema (General disorders) | 95/302 (95) | 101/319 (101) | 101/306 (101) | 43/149 (43)
Injection Site Swelling (General disorders) | 74/310 (74) | 86/336 (86) | 80/329 (80) | 35/156 (35)
Irritability (General disorders) | 188/323 (188) | 198/336 (198) | 193/329 (193) | 83/156 (83)
Pyrexia (General disorders) | 75/310 (75) | 85/317 (85) | 85/315 (85) | 32/153 (32)
Anorexia (Metabolism and nutrition disorders) | 62/323 (62) | 75/336 (75) | 70/329 (70) | 29/149 (29)
Somnolence (Nervous system disorders) | 93/323 (93) | 110/336 (110) | 102/329 (102) | 45/156 (45)
Crying (Psychiatric disorders) | 160/323 (160) | 156/336 (156) | 148/329 (148) | 62/156 (62)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications